CLINICAL TRIAL: NCT03347422
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Sutimlimab in Patients With Primary Cold Agglutinin Disease Without a Recent History of Blood Transfusion
Brief Title: A Study to Assess the Efficacy and Safety of BIVV009 (Sutimlimab) in Participants With Primary Cold Agglutinin Disease Without A Recent History of Blood Transfusion
Acronym: Cadenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC16216; 2017-003539-12 (EudraCT Number); BIVV009-04 (Other: Bioverativ Therapeutics Inc.)
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Cold Agglutinin Disease
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — sutimlimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIVV009/BIVV009 (Experimental): Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an intravenous (IV) infusion of BIVV009 6.5 g (for participants less than [<]75 kilograms [kg]) or 7.5 g dose (for participants greater than or equal to [>=]75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26), received placebo on Week 26 and continued to receive BIVV009 6.5 or 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks (for 6.5 g) or 121 weeks (for 7.5 g). All participants who completed Part A elected to continue in Part B.
  Interventions: Drug: sutimlimab (BIVV009)
- Placebo/BIVV009 (Experimental): Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of placebo matched to BIVV009 on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26) received BIVV009 6.5 (if <75 kg) or 7.5 g (if >=75 kg) in Part B, on Week 26 and Week 27 and every 2 weeks thereafter for up to an additional 123 weeks (for 6.5 g) or 137 weeks (for 7.5 g). All participants who completed Part A elected to continue in Part B.
  Interventions: Drug: sutimlimab (BIVV009); Drug: placebo

INTERVENTIONS:
Drug: sutimlimab (BIVV009) — Pharmaceutical form: solution for injection Route of administration: intravenous (i.v.)
Drug: placebo — Pharmaceutical form: solution for injection Route of administration: intravenous (i.v.)
  Arms: Placebo/BIVV009

SUMMARY:
The purpose of Part A was to determine whether sutimlimab administration resulted in a greater than or equal to (>=)1.5 grams per deciliter (g/dL) increase in hemoglobin (Hgb) level and avoidance of transfusion in participants with primary cold agglutinin disease (CAD) without a recent history of blood transfusion. The purpose of Part B was to evaluate the long-term safety and tolerability of sutimlimab in participants with primary CAD.

DETAILED DESCRIPTION:
The planned total study duration per participant was approximately 1.5 to 2.5 years.

ELIGIBILITY:
Inclusion criteria:

* Body weight of >=39 kg at screening.
* Confirmed diagnosis of primary CAD based on the following criteria: a) Chronic hemolysis, b) Polyspecific direct antiglobulin test (DAT) positive, c) Monospecific DAT strongly positive for C3d, d) Cold agglutinin titer >= 64 at 4 degree Celsius, and e) Immunoglobulin G DAT less than or equal to (<=) 1+, and, f) No overt malignant disease.
* Hemoglobin level <= 10.0 g/dL.
* Bilirubin level above the normal reference range, including participants with Gilbert's Syndrome.

Exclusion criteria:

* Cold agglutinin syndrome secondary to infection, rheumatologic disease, or active hematologic malignancy.
* History of blood transfusion within 6 months of screening, or history of more than one blood transfusion within 12 months of screening.
* Clinically relevant infection of any kind within the month preceding enrollment (example, active hepatitis C, pneumonia).
* Clinical diagnosis of systemic lupus erythematosus; or other autoimmune disorders with anti-nuclear antibodies at screening. Anti-nuclear antibodies of long-standing duration without associated clinical symptoms would be adjudicated on a case-by-case basis during the confirmatory review of participant eligibility.
* Positive hepatitis panel (including hepatitis B surface antigen and/or hepatitis C virus antibody) prior to or at screening.
* Positive human immunodeficiency virus antibody at screening.
* Treatment with rituximab monotherapy within 3 months or rituximab combination therapies (example, with bendamustine, fludarabine, ibrutinib, or cytotoxic drugs) within 6 months prior to enrollment.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (53):
- United States (14):
  - Arizona Oncology Associates PC, Tucson, Arizona
  - USC/Keck School of Medicine, Los Angeles, California
  - Georgetown University Medical Center, Georgetown, District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, New York, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - East Carolina University, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UW Hospitals and Clinics, Madison, Wisconsin
- Australia (4):
  - USC Health Clinics, Buderim, Queensland
  - Ballarat Oncology & Haematology, Ballarat, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Perth Blood Institute, West Perth, Western Australia
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - ZNA Stuivenberg, Antwerp
  - University Hospitals Leuven, Leuven
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- France (4):
  - CHU d'Angers, Angers
  - Hôpital de Caen, Caen
  - Centre Hospitalier Henri Mondor, Créteil
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - Universitätsklinikum Essen, Essen
  - Univ Ulm, Inst Klin. Transfusions. Immungen, Ulm
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Laniado Hospital, Netanya
- Italy (4):
  - A. O. Spedali Civili di Brescia, Brescia
  - Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - U.O.C. Ematologia- Policlinico "A. Gemelli", Rome
  - U.O.C. Ematologia Ospedale San Bortolo, Vicenza
- Japan (6):
  - Japanese Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Aichi Medical University Hospital, Nagakute
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
- Norway (2):
  - Haukeland University Hospital, Bergen
  - St Olavs Hospital, Avdeling for blodsykdommer, Trondheim
- Spain (4):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clinci i Provincial de Barcelona, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Dr. Peset, Valencia
- United Kingdom (3):
  - St James Hospital, Leeds, Leeds
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Roth A, Broome CM, Barcellini W, Jilma B, Hill QA, Cella D, Tvedt THA, Yamaguchi M, Lee M, Shafer F, Wardecki M, Jiang X, Patel P, Joly F, Weitz IC. Sutimlimab provides clinically meaningful improvements in patient-reported outcomes in patients with cold agglutinin disease: Results from the randomised, placebo-controlled, Phase 3 CADENZA study. Eur J Haematol. 2023 Mar;110(3):280-288. doi: 10.1111/ejh.13903. Epub 2022 Dec 9. PMID 36403132
- [Derived] Roth A, Berentsen S, Barcellini W, D'Sa S, Jilma B, Michel M, Weitz IC, Yamaguchi M, Nishimura JI, Vos JMI, Storek M, Wong N, Patel P, Jiang X, Vagge DS, Wardecki M, Shafer F, Lee M, Broome CM. Sutimlimab in patients with cold agglutinin disease: results of the randomized placebo-controlled phase 3 CADENZA trial. Blood. 2022 Sep 1;140(9):980-991. doi: 10.1182/blood.2021014955. PMID 35687757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 sites in 13 countries. Out of 66 screened participants, a total of 42 participants were enrolled and randomized from 17 March 2018 to 30 March 2020. This study consisted of 2 Parts: Part A and Part B.
Pre-assignment Details: Participants were stratified based on baseline body weight to receive BIVV009 6.5 grams (g) (if <75 kg) or 7.5 g (if >=75 kg). As planned, data presented as: 1) Dose-wise (2 dose cohorts: BIVV009 6.5 g & BIVV009 7.5 g) for safety outcome measures and adverse events (AEs). 2) combined population (BIVV009 at any dose) for efficacy outcome measures.
Groups:
- BIVV009/BIVV009: Participants with primary Cold Agglutinin Disease (CAD) and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an intravenous (IV) infusion of BIVV009 6.5 g (for participants less than [<]75 kilograms [kg]) or 7.5 g dose (for participants greater than or equal to [>=]75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26), received placebo on Week 26 and continued to receive BIVV009 6.5 or 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks (for 6.5 g) or 121 weeks (for 7.5 g). All participants who completed Part A elected to continue in Part B.
Period: Part A (26 Weeks)
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Started | 22 | 20
Completed | 19 | 20
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Part B (149 Weeks)
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Started | 19 | 20
Completed | 16 | 16
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) which included all randomized participants who received at least 1 dose (including partial dose) of study drug (BIVV009 or placebo).
Groups:
- BIVV009/BIVV009: Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of BIVV009 6.5 g (for participants <75 kg) or 7.5 g dose (for participants >=75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25. Participants who completed Part A per protocol through the end of treatment visit (Week 26), received placebo on Week 26 and continued to receive BIVV009 6.5 or 7.5 g in Part B, every 2 weeks starting at Week 27 for up to an additional 149 weeks (for 6.5 g) or 121 weeks (for 7.5 g). All participants who completed Part A elected to continue in Part B.
- Total: Total of all reporting groups
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009 | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.9) | 68.2 (10.1) | 66.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants With Response to Treatment
Description: A participant was considered a responder: if he or she did not receive blood transfusion from Week 5 through Week 26 (end of treatment) and did not receive treatment for CAD beyond what was permitted per protocol. Additionally, participant's hemoglobin (Hgb) level must have increased to >=1.5 grams per deciliter (g/dL) from baseline (defined as last Hgb value before administration of first dose of study drug) at treatment assessment timepoint (defined as average of values from the Week 23, 25, and 26 visits). Percentage of responders was calculated together with 95% exact Clopper-Pearson confidence interval (CI).
Time Frame: From Week 5 through Week 26
Population: Analysis was performed on Part A-full analysis set (FAS) which included all randomized participants who received at least 1 dose (including partial dose) of study drug (BIVV009 or placebo). Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either at 6.5 or 7.5 g] and placebo in Part A.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BIVV009: Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of BIVV009 6.5 g (for participants <75 kg) or 7.5 g dose (for participants >=75 kg) on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
- Placebo: Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of placebo matched to BIVV009 on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 22 | 20
percentage of participants | 72.7 [49.8 to 89.3] | 15.0 [3.2 to 37.9]
Statistical Analysis 1: Comparison: BIVV009 vs Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when primary outcome measure was statistically significant at two-sided 0.05 level; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance was 0.05; Odds Ratio (OR) = 15.94, 95% CI 2-sided [2.88 to 88.04] — Stratified by baseline hemoglobin (< median versus >=median) and geographic region (Asia/Other, North America, and Europe)

2. Primary Outcome: Part B: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Adverse Event (AE): any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Treatment emergent serious adverse events (TESAEs) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect, was medically important event. Treatment emergent adverse events (TEAEs): AEs that developed, worsened or became serious during the treatment-emergent (TE) period (from first investigational medicinal product [IMP] administration in Part B to last IMP administration + 9 weeks follow-up period).
Time Frame: Part B, 6.5 g cohort: From first dose (Week 26) up to 149 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 184); Part B, 7.5 g cohort: From first dose (Week 26) up to 137 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 172)
Population: Analyzed on Part B safety analysis set (SAS) which included all participants who received at least 1 dose (including partial dose) of study drug in Part B. Data for this outcome measures was planned to be collected and analyzed separately for each dose of BIVV009 (6.5 g and 7.5 g).
Measure: Count of Participants; unit: Participants
Groups:
- Part B: BIVV009 6.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) were eligible to be enrolled in Part B where they were treated for up to an additional 149 weeks. Participants who received placebo in Part A received BIVV009 6.5 g on Week 26, Week 27 and every 2 weeks thereafter; participants who received BIVV009 6.5 g in Part A received placebo on Week 26, BIVV009 6.5 g on Week 27 and every 2 weeks thereafter for up to an additional 149 weeks.
- Part B: BIVV009 7.5 g: Participants who completed Part A per protocol through the end of treatment visit (Week 26) were eligible to be enrolled in Part B where they were treated for up to an additional 137 weeks. Participants who received placebo in Part A received BIVV009 7.5 g on Week 26, Week 27 and every 2 weeks thereafter; participants who received BIVV009 7.5 g in Part A received placebo on Week 26, BIVV009 7.5 g on Week 27 and every 2 weeks thereafter for up to an additional 137 weeks.
Arm/Group | Part B: BIVV009 6.5 g | Part B: BIVV009 7.5 g
Number analyzed (Participants) | 32 | 7
Participants
  TEAEs | 29 | 7
  TESAEs | 6 | 1

3. Secondary Outcome: Part A: Mean Change From Baseline in Hemoglobin (Hgb) Level at the Treatment Assessment Timepoint
Description: Mean change from baseline (Week 0) in Hemoglobin (Hgb) at the treatment assessment timepoint is reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. Least squares (LS) mean and 95 % confidence interval (CI) was assessed by Mixed Model for Repeated Measures (MMRM) approach using heterogeneous Toeplitz (TOEPH) covariance matrix with change from baseline as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline (Week 0), treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: Analysis was performed on Part A-FAS. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either at 6.5 or 7.5 g] and placebo in Part A.
Measure: Least Squares Mean (95% Confidence Interval); unit: grams per deciliter
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 22 | 20
grams per deciliter | 2.66 [2.09 to 3.22] | 0.09 [-0.50 to 0.68]
Statistical Analysis 1: Comparison: BIVV009 vs Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.05 level; Test type: Superiority; p < 0.001, Mixed model for repeated measures — Threshold of significance at 0.05 level; LS mean difference = 2.56, 95% CI 2-sided [1.75 to 3.38], Standard Error of Mean 0.408

4. Secondary Outcome: Part A: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score at the Treatment Assessment Timepoint
Description: FACIT-Fatigue scale consists of 13 questions assessed using a 5-point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). Responses to each question were added to obtain a total score. Total score ranged from 0 to 52, with higher score indicating more fatigue. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. LS mean and 95% CI was assessed by MMRM approach using TOEPH covariance matrix with change from baseline (Week 0) as the dependent variable and baseline value and visits as independent variables. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline (Week 0), treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: Analysis was performed on Part A-FAS. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]) and placebo in Part A.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 22 | 20
score on a scale | 10.83 [7.45 to 14.22] | 1.91 [-1.65 to 5.46]
Statistical Analysis 1: Comparison: BIVV009 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, Mixed model for repeated measures — Threshold of significance at 0.05 level; LS mean difference = 8.93, 95% CI 2-sided [4.00 to 13.85], Standard Error of Mean 2.450

5. Secondary Outcome: Part A: Mean Change From Baseline in Total Bilirubin Levels at the Treatment Assessment Timepoint
Description: Mean change from baseline (Week 0) in total bilirubin at the treatment assessment timepoint is reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline (Week 0), treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: Analysis was performed on Part A-FAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either at 6.5 or 7.5 g] and placebo in Part A.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 19 | 20
micromoles per liter | -22.881 (10.401) | -1.388 (13.901)

6. Secondary Outcome: Part A: Mean Change From Baseline in Lactate Dehydrogenase (LDH) at the Treatment Assessment Timepoint
Description: Mean change from baseline (Week 0) in LDH at the treatment assessment timepoint is reported in this outcome measure. Treatment assessment timepoint was defined as the average of the values from the Week 23, 25, and 26 visits. Baseline was defined as the last non-missing value prior to the first administration of study drug.
Time Frame: Baseline (Week 0), treatment assessment timepoint (i.e., average of Week 23, 25 and 26)
Population: Analysis was performed on Part A-FAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]) and placebo in Part A.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 19 | 20
units per liter | -150.833 (160.824) | 7.600 (212.690)

7. Secondary Outcome: Part A: Percentage of Participants With Solicited Symptomatic Anemia at Week 26
Description: Symptomatic anemia was defined as having following symptoms: i. Fatigue; ii. Weakness; iii. Shortness of breath; iv. Palpitations, fast heartbeat; v. Light headedness and/or vi. Chest pain. Percentage of participants with solicited symptomatic anemia symptoms was reported in this outcome measure.
Time Frame: Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | BIVV009 | Placebo
Number analyzed (Participants) | 19 | 19
percentage of participants
  Fatigue | 31.6 | 68.4
  Weakness | 5.3 | 31.6
  Shortness of breath | 5.3 | 36.8
  Palpitations | 0 | 15.8
  Light headedness | 5.3 | 15.8
  Chest pain | 0 | 5.3

8. Secondary Outcome: Part B: Change From Baseline in Hemoglobin (Hgb) Level at Each Specified Time Points
Description: Change from baseline (Week 0) in Hgb levels at each specified time points (i.e., Week 27, 29, 31, 33, 35, 37, 39, 41, 43,45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 81, 83,85,87, 89,91, 93, 95, 97, 99,101,103, 105, 107,109, 111,113,115,117,119, 121,123, 125, 127,129,131,133,135,137,139,141,143,145,147,149,151,153, 155,157,159,161,163,165,167,169,171,173,175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. Early Termination (ET) visit/safety follow up (SFU) visit was 9 weeks after administration of last dose (i.e., up to Week 184). Here, "0" in the number analyzed field signifies that none of participants were available for assessment at the specified timepoints.
Time Frame: Baseline (Week 0), every 2 weeks starting from Week 27 till Week 175 and at ET/SFU visit (i.e., up to Week 184)
Population: Analyzed on Part B-FAS which included all participants who enrolled in Part B and received at least 1 dose (including partial dose) of study drug (BIVV009). Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
grams per deciliter
  Week 27 | 2.647 (1.348) | 1.125 (1.545)
  Week 29: number analyzed (Participants) | 17 | 18
  Week 29 | 2.507 (1.669) | 1.947 (1.467)
  Week 31: number analyzed (Participants) | 18 | 19
  Week 31 | 2.490 (1.550) | 2.358 (1.471)
  Week 33: number analyzed (Participants) | 18 | 19
  Week 33 | 2.519 (1.520) | 1.987 (2.054)
  Week 35: number analyzed (Participants) | 17 | 19
  Week 35 | 2.611 (1.522) | 1.977 (2.010)
  Week 37: number analyzed (Participants) | 18 | 19
  Week 37 | 2.197 (1.461) | 2.469 (1.550)
  Week 39: number analyzed (Participants) | 17 | 18
  Week 39 | 2.528 (1.607) | 2.368 (1.835)
  Week 41: number analyzed (Participants) | 19 | 19
  Week 41 | 2.162 (1.636) | 2.074 (1.825)
  Week 43: number analyzed (Participants) | 17 | 19
  Week 43 | 2.436 (1.103) | 2.182 (1.643)
  Week 45: number analyzed (Participants) | 18 | 20
  Week 45 | 2.644 (1.688) | 2.249 (1.858)
  Week 47: number analyzed (Participants) | 16 | 19
  Week 47 | 2.335 (1.108) | 2.315 (2.129)
  Week 49: number analyzed (Participants) | 16 | 18
  Week 49 | 2.531 (1.280) | 2.121 (1.883)
  Week 51: number analyzed (Participants) | 16 | 19
  Week 51 | 2.349 (1.260) | 2.394 (1.870)
  Week 53: number analyzed (Participants) | 16 | 18
  Week 53 | 2.346 (1.182) | 2.411 (1.786)
  Week 55: number analyzed (Participants) | 17 | 18
  Week 55 | 2.438 (1.396) | 2.539 (1.403)
  Week 57: number analyzed (Participants) | 16 | 17
  Week 57 | 2.531 (1.446) | 2.250 (1.774)
  Week 59: number analyzed (Participants) | 17 | 17
  Week 59 | 2.590 (1.397) | 2.008 (2.615)
  Week 61: number analyzed (Participants) | 17 | 18
  Week 61 | 4.073 (6.761) | 2.059 (1.911)
  Week 63: number analyzed (Participants) | 17 | 17
  Week 63 | 2.382 (1.546) | 2.102 (1.780)
  Week 65: number analyzed (Participants) | 16 | 17
  Week 65 | 2.925 (1.447) | 2.311 (1.986)
  Week 67: number analyzed (Participants) | 17 | 17
  Week 67 | 4.170 (6.509) | 2.534 (2.036)
  Week 69: number analyzed (Participants) | 16 | 17
  Week 69 | 2.777 (1.411) | 2.505 (2.093)
  Week 71: number analyzed (Participants) | 14 | 15
  Week 71 | 2.654 (1.495) | 2.357 (1.758)
  Week 73: number analyzed (Participants) | 15 | 16
  Week 73 | 2.800 (2.132) | 2.197 (1.989)
  Week 75: number analyzed (Participants) | 15 | 16
  Week 75 | 2.391 (1.700) | 2.175 (2.151)
  Week 77: number analyzed (Participants) | 14 | 16
  Week 77 | 3.074 (2.088) | 2.451 (1.878)
  Week 79: number analyzed (Participants) | 13 | 15
  Week 79 | 2.614 (1.874) | 2.419 (2.247)
  Week 81: number analyzed (Participants) | 14 | 17
  Week 81 | 2.598 (1.801) | 2.458 (1.579)
  Week 83: number analyzed (Participants) | 14 | 13
  Week 83 | 2.469 (1.777) | 2.762 (1.539)
  Week 85: number analyzed (Participants) | 12 | 15
  Week 85 | 2.755 (1.942) | 2.489 (1.375)
  Week 87: number analyzed (Participants) | 13 | 15
  Week 87 | 2.477 (1.779) | 2.765 (1.605)
  Week 89: number analyzed (Participants) | 12 | 13
  Week 89 | 2.551 (1.835) | 2.482 (2.004)
  Week 91: number analyzed (Participants) | 11 | 12
  Week 91 | 2.380 (2.084) | 2.556 (1.538)
  Week 93: number analyzed (Participants) | 11 | 12
  Week 93 | 2.931 (2.386) | 2.655 (2.033)
  Week 95: number analyzed (Participants) | 11 | 12
  Week 95 | 2.262 (2.014) | 2.578 (1.970)
  Week 97: number analyzed (Participants) | 11 | 12
  Week 97 | 2.413 (2.262) | 2.551 (1.544)
  Week 99: number analyzed (Participants) | 11 | 13
  Week 99 | 2.019 (1.799) | 2.412 (1.822)
  Week 101: number analyzed (Participants) | 11 | 12
  Week 101 | 2.276 (1.986) | 2.171 (1.852)
  Week 103: number analyzed (Participants) | 11 | 13
  Week 103 | 2.378 (2.342) | 2.527 (1.807)
  Week 105: number analyzed (Participants) | 11 | 12
  Week 105 | 2.291 (1.719) | 2.321 (1.805)
  Week 107: number analyzed (Participants) | 11 | 13
  Week 107 | 2.319 (1.511) | 2.560 (1.858)
  Week 109: number analyzed (Participants) | 11 | 11
  Week 109 | 2.509 (1.772) | 2.645 (1.608)
  Week 111: number analyzed (Participants) | 11 | 12
  Week 111 | 2.416 (1.908) | 2.750 (1.707)
  Week 113: number analyzed (Participants) | 11 | 12
  Week 113 | 2.860 (1.832) | 2.268 (1.497)
  Week 115: number analyzed (Participants) | 10 | 10
  Week 115 | 2.622 (1.986) | 2.326 (1.809)
  Week 117: number analyzed (Participants) | 9 | 11
  Week 117 | 3.135 (1.598) | 2.474 (1.808)
  Week 119: number analyzed (Participants) | 9 | 10
  Week 119 | 3.106 (1.493) | 2.608 (2.045)
  Week 121: number analyzed (Participants) | 9 | 8
  Week 121 | 3.388 (1.616) | 2.325 (2.223)
  Week 123: number analyzed (Participants) | 9 | 9
  Week 123 | 3.255 (1.346) | 2.878 (2.667)
  Week 125: number analyzed (Participants) | 8 | 7
  Week 125 | 3.197 (1.366) | 1.700 (2.684)
  Week 127: number analyzed (Participants) | 7 | 8
  Week 127 | 3.371 (1.551) | 2.102 (3.211)
  Week 129: number analyzed (Participants) | 7 | 7
  Week 129 | 3.171 (1.566) | 2.129 (2.739)
  Week 131: number analyzed (Participants) | 6 | 6
  Week 131 | 3.453 (1.823) | 1.423 (3.184)
  Week 133: number analyzed (Participants) | 5 | 4
  Week 133 | 3.520 (1.707) | 2.025 (1.167)
  Week 135: number analyzed (Participants) | 5 | 5
  Week 135 | 3.611 (1.458) | 3.048 (1.620)
  Week 137: number analyzed (Participants) | 4 | 3
  Week 137 | 4.074 (2.392) | 2.400 (1.808)
  Week 139: number analyzed (Participants) | 5 | 3
  Week 139 | 3.929 (1.889) | 3.334 (2.669)
  Week 141: number analyzed (Participants) | 3 | 3
  Week 141 | 3.500 (0.656) | 2.733 (1.674)
  Week 143: number analyzed (Participants) | 4 | 3
  Week 143 | 3.220 (1.064) | 2.985 (1.904)
  Week 145: number analyzed (Participants) | 2 | 3
  Week 145 | 3.350 (0.636) | 3.467 (2.108)
  Week 147: number analyzed (Participants) | 3 | 2
  Week 147 | 3.202 (0.591) | 2.300 (0.566)
  Week 149: number analyzed (Participants) | 1 | 2
  Week 149 | 2.900 | 2.550 (0.778)
  Week 151: number analyzed (Participants) | 2 | 1
  Week 151 | 2.961 (0.370) | 3.000
  Week 153: number analyzed (Participants) | 1 | 1
  Week 153 | 2.800 | 2.800
  Week 155: number analyzed (Participants) | 1 | 1
  Week 155 | 2.700 | 3.600
  Week 157: number analyzed (Participants) | 1 | 1
  Week 157 | 2.700 | 3.000
  Week 159: number analyzed (Participants) | 1 | 1
  Week 159 | 3.300 | 2.300
  Week 161: number analyzed (Participants) | 1 | 1
  Week 161 | 4.100 | 2.400
  Week 163: number analyzed (Participants) | 1 | 1
  Week 163 | 4.100 | 2.600
  Week 165: number analyzed (Participants) | 1 | 0
  Week 165 | 3.800 |
  Week 167: number analyzed (Participants) | 1 | 0
  Week 167 | 4.700 |
  Week 169: number analyzed (Participants) | 1 | 0
  Week 169 | 4.300 |
  Week 171: number analyzed (Participants) | 1 | 0
  Week 171 | 4.200 |
  Week 173: number analyzed (Participants) | 1 | 0
  Week 173 | 4.000 |
  Week 175: number analyzed (Participants) | 1 | 0
  Week 175 | 2.500 |
  ET/SFU Visit: number analyzed (Participants) | 17 | 18
  ET/SFU Visit | 0.149 (2.073) | 0.359 (1.872)

9. Secondary Outcome: Part B: Change From Baseline in Total Bilirubin Levels at Each Specified Time Points
Description: Change from baseline (Week 0) in total bilirubin levels at each specified time points (i.e., Week 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65,67,69,71,73,75, 77, 79, 81,83, 85, 87, 89, 91, 93, 95, 97, 99,101,103, 105, 107,109, 111,113,115,117,119, 121, 123, 125, 127,129,131,133,135,137,139,141,143, 145,147,149,151,153,155,157,159, 161,163,165,167,169,171,173,175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184). Here, "0" in the number analyzed field signifies that none of participants were available for assessment at the specified timepoints.
Time Frame: Baseline (Week 0), every 2 weeks starting from Week 27 till Week 175 and at ET/SFU visit (i.e., up to Week 184)
Population: Analysis was performed on Part B-FAS. Here, 'overall number of participants analyzed'=participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 17 | 18
micromoles per liter
  Week 27 | -22.965 (9.899) | -18.761 (13.353)
  Week 29: number analyzed (Participants) | 16 | 18
  Week 29 | -20.119 (12.170) | -19.889 (14.500)
  Week 31: number analyzed (Participants) | 16 | 17
  Week 31 | -21.675 (11.025) | -22.153 (14.962)
  Week 33: number analyzed (Participants) | 15 | 16
  Week 33 | -19.860 (11.527) | -24.263 (15.169)
  Week 35: number analyzed (Participants) | 15 | 16
  Week 35 | -20.540 (10.557) | -21.888 (13.930)
  Week 37: number analyzed (Participants) | 16 | 15
  Week 37 | -21.350 (13.234) | -22.527 (16.315)
  Week 39: number analyzed (Participants) | 15 | 15
  Week 39 | -23.493 (11.425) | -21.173 (15.901)
  Week 41: number analyzed (Participants) | 16 | 16
  Week 41 | -18.694 (12.189) | -21.138 (16.150)
  Week 43: number analyzed (Participants) | 15 | 16
  Week 43 | -20.593 (11.449) | -21.544 (16.603)
  Week 45: number analyzed (Participants) | 16 | 18
  Week 45 | -18.556 (11.213) | -20.156 (16.757)
  Week 47: number analyzed (Participants) | 14 | 18
  Week 47 | -20.400 (9.803) | -20.250 (15.536)
  Week 49: number analyzed (Participants) | 14 | 17
  Week 49 | -21.450 (10.271) | -21.024 (13.630)
  Week 51: number analyzed (Participants) | 14 | 16
  Week 51 | -19.686 (11.072) | -19.444 (15.942)
  Week 53: number analyzed (Participants) | 15 | 17
  Week 53 | -19.107 (11.267) | -20.335 (17.126)
  Week 55: number analyzed (Participants) | 13 | 16
  Week 55 | -19.354 (12.209) | -23.481 (12.300)
  Week 57: number analyzed (Participants) | 13 | 15
  Week 57 | -21.708 (10.467) | -18.953 (15.825)
  Week 59: number analyzed (Participants) | 14 | 15
  Week 59 | -19.979 (9.706) | -19.820 (16.209)
  Week 61: number analyzed (Participants) | 13 | 15
  Week 61 | -18.254 (10.541) | -21.073 (17.457)
  Week 63: number analyzed (Participants) | 15 | 15
  Week 63 | -21.587 (9.680) | -21.753 (16.663)
  Week 65: number analyzed (Participants) | 14 | 14
  Week 65 | -20.400 (9.866) | -20.950 (19.833)
  Week 67: number analyzed (Participants) | 15 | 14
  Week 67 | -22.680 (10.317) | -20.150 (20.250)
  Week 69: number analyzed (Participants) | 14 | 15
  Week 69 | -21.279 (9.423) | -17.827 (22.194)
  Week 71: number analyzed (Participants) | 12 | 13
  Week 71 | -19.008 (8.255) | -20.585 (21.125)
  Week 73: number analyzed (Participants) | 12 | 15
  Week 73 | -23.058 (7.766) | -20.080 (17.803)
  Week 75: number analyzed (Participants) | 12 | 14
  Week 75 | -21.492 (7.453) | -20.771 (20.261)
  Week 77: number analyzed (Participants) | 12 | 14
  Week 77 | -23.267 (8.972) | -19.814 (19.337)
  Week 79: number analyzed (Participants) | 12 | 15
  Week 79 | -21.125 (12.701) | -21.027 (19.830)
  Week 81: number analyzed (Participants) | 11 | 13
  Week 81 | -19.255 (9.478) | -22.331 (20.117)
  Week 83: number analyzed (Participants) | 12 | 11
  Week 83 | -16.567 (12.565) | -25.091 (13.838)
  Week 85: number analyzed (Participants) | 11 | 13
  Week 85 | -18.045 (12.183) | -23.292 (12.976)
  Week 87: number analyzed (Participants) | 10 | 11
  Week 87 | -19.990 (12.043) | -21.473 (14.444)
  Week 89: number analyzed (Participants) | 10 | 11
  Week 89 | -17.790 (11.036) | -24.782 (13.390)
  Week 91: number analyzed (Participants) | 9 | 11
  Week 91 | -16.944 (13.476) | -23.091 (14.949)
  Week 93: number analyzed (Participants) | 9 | 10
  Week 93 | -18.300 (11.132) | -24.970 (13.852)
  Week 95: number analyzed (Participants) | 8 | 11
  Week 95 | -18.613 (12.265) | -23.564 (11.122)
  Week 97: number analyzed (Participants) | 9 | 9
  Week 97 | -18.656 (11.462) | -26.122 (11.870)
  Week 99: number analyzed (Participants) | 9 | 11
  Week 99 | -17.389 (10.932) | -23.700 (12.919)
  Week 101: number analyzed (Participants) | 9 | 10
  Week 101 | -18.411 (10.175) | -25.940 (12.309)
  Week 103: number analyzed (Participants) | 9 | 11
  Week 103 | -18.178 (11.156) | -22.655 (11.308)
  Week 105: number analyzed (Participants) | 9 | 10
  Week 105 | -19.422 (8.444) | -26.920 (10.996)
  Week 107: number analyzed (Participants) | 9 | 11
  Week 107 | -18.100 (9.955) | -23.018 (12.755)
  Week 109: number analyzed (Participants) | 9 | 9
  Week 109 | -18.456 (10.606) | -25.422 (14.100)
  Week 111: number analyzed (Participants) | 9 | 10
  Week 111 | -19.767 (9.992) | -24.380 (12.298)
  Week 113: number analyzed (Participants) | 9 | 10
  Week 113 | -19.389 (9.192) | -23.940 (15.514)
  Week 115: number analyzed (Participants) | 9 | 9
  Week 115 | -19.622 (8.194) | -21.533 (14.215)
  Week 117: number analyzed (Participants) | 8 | 8
  Week 117 | -22.088 (10.247) | -22.225 (15.256)
  Week 119: number analyzed (Participants) | 8 | 8
  Week 119 | -20.038 (8.529) | -22.713 (14.859)
  Week 121: number analyzed (Participants) | 8 | 6
  Week 121 | -22.063 (7.215) | -21.183 (10.750)
  Week 123: number analyzed (Participants) | 8 | 7
  Week 123 | -21.438 (8.058) | -22.029 (12.421)
  Week 125: number analyzed (Participants) | 7 | 5
  Week 125 | -20.657 (8.889) | -19.560 (12.997)
  Week 127: number analyzed (Participants) | 6 | 6
  Week 127 | -20.550 (9.782) | -21.433 (15.850)
  Week 129: number analyzed (Participants) | 6 | 5
  Week 129 | -22.883 (11.291) | -19.020 (11.749)
  Week 131: number analyzed (Participants) | 5 | 5
  Week 131 | -19.420 (12.936) | -23.100 (15.797)
  Week 133: number analyzed (Participants) | 4 | 4
  Week 133 | -27.600 (7.477) | -17.450 (16.917)
  Week 135: number analyzed (Participants) | 4 | 5
  Week 135 | -29.500 (7.816) | -21.900 (19.552)
  Week 137: number analyzed (Participants) | 3 | 2
  Week 137 | -28.833 (8.615) | -11.650 (18.173)
  Week 139: number analyzed (Participants) | 4 | 3
  Week 139 | -25.800 (9.081) | -24.733 (17.470)
  Week 141: number analyzed (Participants) | 2 | 3
  Week 141 | -34.400 (2.404) | -13.833 (16.669)
  Week 143: number analyzed (Participants) | 3 | 3
  Week 143 | -26.967 (9.235) | -20.033 (22.861)
  Week 145: number analyzed (Participants) | 2 | 3
  Week 145 | -32.900 (3.677) | -18.100 (27.217)
  Week 147: number analyzed (Participants) | 3 | 2
  Week 147 | -29.300 (7.418) | -3.300 (34.083)
  Week 149: number analyzed (Participants) | 1 | 2
  Week 149 | -31.700 | -7.300 (28.284)
  Week 151: number analyzed (Participants) | 2 | 1
  Week 151 | -21.500 (0.566) | 0.300
  Week 153: number analyzed (Participants) | 1 | 1
  Week 153 | -30.800 | -11.400
  Week 155: number analyzed (Participants) | 1 | 1
  Week 155 | -35.300 | 0.700
  Week 157: number analyzed (Participants) | 1 | 1
  Week 157 | -32.400 | -0.100
  Week 159: number analyzed (Participants) | 1 | 1
  Week 159 | -32.500 | 4.700
  Week 161: number analyzed (Participants) | 1 | 1
  Week 161 | -36.800 | 5.500
  Week 163: number analyzed (Participants) | 1 | 1
  Week 163 | -37.100 | 13.000
  Week 165: number analyzed (Participants) | 1 | 0
  Week 165 | -36.300 |
  Week 167: number analyzed (Participants) | 1 | 0
  Week 167 | -34.300 |
  Week 169: number analyzed (Participants) | 1 | 0
  Week 169 | -32.700 |
  Week 171: number analyzed (Participants) | 1 | 0
  Week 171 | -33.100 |
  Week 173: number analyzed (Participants) | 1 | 0
  Week 173 | -32.100 |
  Week 175: number analyzed (Participants) | 1 | 0
  Week 175 | -28.400 |
  ET/SFU Visit: number analyzed (Participants) | 17 | 17
  ET/SFU Visit | 1.976 (9.444) | 1.165 (18.773)

10. Secondary Outcome: Part B: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score (Quality of Life) at Each Specified Time Points
Description: FACIT-Fatigue scale consists of 13 questions assessed using a 5-point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). Responses to each question were added to obtain a total score. The Total score ranged from 0 to 52, with higher score indicating more fatigue. Baseline (Week 0) was defined as the last non-missing value prior to the first administration of study drug in Part A. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: Baseline (Week 0), Weeks 39, 51, 63, 75, 87, 99, 111, 123, 135, 147, 159, 171 and ET Visit/SFU visit (i.e., up to Week 184)
Population: Analysis was performed on Part B-FAS. Here, 'number analyzed'=participants with available data for each specified category and "0" in the number analyzed field signifies that none of participants were available for assessment at the specified timepoints. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
score on a scale
  Week 39: number analyzed (Participants) | 18 | 18
  Week 39 | 11.048 (12.333) | 7.958 (12.003)
  Week 51: number analyzed (Participants) | 15 | 16
  Week 51 | 10.080 (11.506) | 6.354 (9.680)
  Week 63: number analyzed (Participants) | 16 | 16
  Week 63 | 10.672 (13.225) | 8.499 (11.146)
  Week 75: number analyzed (Participants) | 13 | 14
  Week 75 | 9.861 (12.953) | 10.304 (9.722)
  Week 87: number analyzed (Participants) | 13 | 15
  Week 87 | 11.015 (13.972) | 8.483 (11.323)
  Week 99: number analyzed (Participants) | 11 | 13
  Week 99 | 12.109 (14.786) | 8.788 (10.985)
  Week 111: number analyzed (Participants) | 11 | 12
  Week 111 | 11.563 (13.411) | 10.688 (11.768)
  Week 123: number analyzed (Participants) | 9 | 9
  Week 123 | 10.806 (13.736) | 6.583 (16.613)
  Week 135: number analyzed (Participants) | 5 | 5
  Week 135 | 16.683 (18.953) | 12.650 (15.243)
  Week 147: number analyzed (Participants) | 2 | 2
  Week 147 | 9.208 (1.120) | 0.500 (2.121)
  Week 159: number analyzed (Participants) | 1 | 1
  Week 159 | 20.000 | 10.000
  Week 171: number analyzed (Participants) | 1 | 0
  Week 171 | 15.000 |
  ET/SFU Visit: number analyzed (Participants) | 19 | 18
  ET/SFU Visit | -1.257 (10.399) | -1.551 (12.840)

11. Secondary Outcome: Part B: Change From Baseline in 12-Item Short-Form Survey (SF-12) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Each Specified Time Points
Description: SF-12: 12 item-questionnaire assessed health-related quality of life (HRQOL), contained 12 items, categorized into 8 domains (subscales) of functioning and well-being: physical functioning, role-physical, role emotional, mental health, bodily pain, general health, vitality and social functioning, with each domain score ranged from 0 (poor health) to 100 (better health). Higher scores = good health condition. These 8 domains were further summarized into 2 summary scores, PCS and MCS that ranged from 0 (poor health) to 100 (better health). Higher scores = better HRQOL. Baseline (Week 0): last non-missing value prior to first administration of study drug in Part A. ET visit/SFU visit: 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
score on a scale
  Week 39-PCS: number analyzed (Participants) | 18 | 18
  Week 39-PCS | 4.814 (8.830) | 6.745 (11.255)
  Week 39-MCS: number analyzed (Participants) | 18 | 18
  Week 39-MCS | 8.543 (9.155) | 1.151 (11.591)
  Week 51-PCS: number analyzed (Participants) | 14 | 16
  Week 51-PCS | 5.320 (6.913) | 5.654 (8.527)
  Week 51-MCS: number analyzed (Participants) | 14 | 16
  Week 51-MCS | 8.461 (6.754) | 1.704 (8.813)
  Week 63-PCS: number analyzed (Participants) | 16 | 16
  Week 63-PCS | 5.840 (6.916) | 6.216 (9.514)
  Week 63-MCS: number analyzed (Participants) | 16 | 16
  Week 63-MCS | 8.117 (9.955) | 1.722 (10.175)
  Week 75-PCS: number analyzed (Participants) | 12 | 15
  Week 75-PCS | 5.723 (7.563) | 7.661 (10.418)
  Week 75-MCS: number analyzed (Participants) | 12 | 15
  Week 75-MCS | 7.932 (9.279) | 3.519 (7.891)
  Week 87-PCS: number analyzed (Participants) | 12 | 15
  Week 87-PCS | 5.226 (8.196) | 8.778 (12.405)
  Week 87-MCS: number analyzed (Participants) | 12 | 15
  Week 87-MCS | 6.058 (10.981) | 2.219 (9.111)
  Week 99-PCS: number analyzed (Participants) | 10 | 13
  Week 99-PCS | 3.945 (7.463) | 8.262 (12.534)
  Week 99-MCS: number analyzed (Participants) | 10 | 13
  Week 99-MCS | 7.136 (11.850) | 4.682 (7.698)
  Week 111-PCS: number analyzed (Participants) | 10 | 12
  Week 111-PCS | 4.800 (7.985) | 8.080 (12.302)
  Week 111-MCS: number analyzed (Participants) | 10 | 12
  Week 111-MCS | 8.705 (7.777) | 4.411 (10.249)
  Week 123-PCS: number analyzed (Participants) | 9 | 9
  Week 123-PCS | 4.147 (7.110) | 7.973 (13.200)
  Week 123-MCS: number analyzed (Participants) | 9 | 9
  Week 123-MCS | 8.650 (8.323) | -2.538 (13.136)
  Week 135-PCS: number analyzed (Participants) | 5 | 4
  Week 135-PCS | 6.660 (9.096) | 6.070 (13.819)
  Week 135-MCS: number analyzed (Participants) | 5 | 4
  Week 135-MCS | 8.860 (9.817) | 2.790 (6.170)
  Week 147-PCS: number analyzed (Participants) | 2 | 2
  Week 147-PCS | -1.655 (3.769) | -3.740 (1.824)
  Week 147-MCS: number analyzed (Participants) | 2 | 2
  Week 147-MCS | 11.220 (6.095) | -1.110 (0.679)
  Week 159-PCS: number analyzed (Participants) | 1 | 1
  Week 159-PCS | 5.620 | -10.410
  Week 159-MCS: number analyzed (Participants) | 1 | 1
  Week 159-MCS | 16.400 | 9.590
  Week 171-PCS: number analyzed (Participants) | 1 | 0
  Week 171-PCS | 11.980 |
  Week 171-MCS: number analyzed (Participants) | 1 | 0
  Week 171-MCS | 0.250 |
  ET/SFU Visit-PCS: number analyzed (Participants) | 18 | 18
  ET/SFU Visit-PCS | -3.478 (10.875) | -0.429 (10.922)
  ET/SFU Visit-MCS: number analyzed (Participants) | 18 | 18
  ET/SFU Visit-MCS | 1.835 (11.882) | -2.137 (10.148)

12. Secondary Outcome: Part B: Change From Baseline in 5-level European Quality of Life 5- Dimensions 5-Level Questionnaire (EQ-5D-5L) Health State Utility Index and VAS Scores at Each Specified Time Points
Description: EQ-5D-5L included 2 components: health state utility index (descriptive system) and Visual Analog Scale (VAS). EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response option: no problem, slight problem, moderate problem, severe problem and extreme problems measured with Likert scale. EQ-5D-5L responses converted into single index utility score between 0 to 1. Higher score=better health. EQ-5D-5L VAS rated participant's current health state on scale from 0 (worst imaginable health) to 100 (best imaginable health). Baseline (Week 0): last non-missing value prior to first administration of study drug in Part A. ET visit/SFU visit: 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
score on a scale
  Week 39-Index score: number analyzed (Participants) | 17 | 18
  Week 39-Index score | 0.020 (0.165) | 0.054 (0.135)
  Week 51-Index score: number analyzed (Participants) | 15 | 16
  Week 51-Index score | 0.075 (0.173) | -0.008 (0.197)
  Week 63-Index score: number analyzed (Participants) | 16 | 16
  Week 63-Index score | 0.060 (0.214) | 0.015 (0.157)
  Week 75-Index score: number analyzed (Participants) | 13 | 15
  Week 75-Index score | -0.004 (0.144) | 0.063 (0.152)
  Week 87-Index score: number analyzed (Participants) | 13 | 15
  Week 87-Index score | -0.034 (0.240) | 0.059 (0.158)
  Week 99-Index score: number analyzed (Participants) | 11 | 13
  Week 99-Index score | -0.058 (0.216) | 0.058 (0.146)
  Week 111-Index score: number analyzed (Participants) | 11 | 12
  Week 111-Index score | -0.033 (0.205) | 0.050 (0.194)
  Week 123-Index score: number analyzed (Participants) | 9 | 9
  Week 123-Index score | -0.020 (0.235) | 0.031 (0.221)
  Week 135-Index score: number analyzed (Participants) | 5 | 5
  Week 135-Index score | 0.008 (0.351) | 0.094 (0.245)
  Week 147-Index score: number analyzed (Participants) | 2 | 2
  Week 147-Index score | 0.054 (0.037) | -0.087 (0.222)
  Week 159-Index score: number analyzed (Participants) | 1 | 1
  Week 159-Index score | 0.174 | 0.087
  Week 171-Index score: number analyzed (Participants) | 1 | 0
  Week 171-Index score | 0.053 |
  ET/SFU Visit-Index score: number analyzed (Participants) | 19 | 18
  ET/SFU Visit-Index score | -0.108 (0.238) | -0.077 (0.169)
  Week 39-VAS: number analyzed (Participants) | 17 | 18
  Week 39-VAS | 20.647 (16.871) | 12.000 (17.146)
  Week 51-VAS: number analyzed (Participants) | 15 | 16
  Week 51-VAS | 14.800 (27.589) | 9.125 (21.112)
  Week 63-VAS: number analyzed (Participants) | 15 | 16
  Week 63-VAS | 19.867 (21.603) | 14.375 (15.573)
  Week 75-VAS: number analyzed (Participants) | 13 | 15
  Week 75-VAS | 16.846 (22.120) | 18.933 (20.243)
  Week 87-VAS: number analyzed (Participants) | 13 | 15
  Week 87-VAS | 14.077 (25.221) | 16.867 (17.912)
  Week 99-VAS: number analyzed (Participants) | 11 | 13
  Week 99-VAS | 19.364 (20.796) | 18.385 (20.706)
  Week 111-VAS: number analyzed (Participants) | 11 | 12
  Week 111-VAS | 18.273 (19.463) | 22.833 (20.621)
  Week 123-VAS: number analyzed (Participants) | 9 | 9
  Week 123-VAS | 21.667 (18.371) | 18.000 (30.389)
  Week 135-VAS: number analyzed (Participants) | 5 | 5
  Week 135-VAS | 26.000 (20.433) | 23.400 (27.574)
  Week 147-VAS: number analyzed (Participants) | 2 | 2
  Week 147-VAS | 17.500 (17.678) | 3.500 (26.163)
  Week 159-VAS: number analyzed (Participants) | 1 | 1
  Week 159-VAS | 40.000 | 27.000
  Week 171-VAS: number analyzed (Participants) | 1 | 0
  Week 171-VAS | 35.000 |
  ET/SFU Visit-VAS: number analyzed (Participants) | 19 | 18
  ET/SFU Visit-VAS | 1.526 (17.976) | -2.056 (14.957)

13. Secondary Outcome: Part B: Number of Participants With Response to Participant's Global Impression of (Fatigue) Severity (PGIS) Questionnaire at Each Specified Time Points
Description: The PGIS is a self-reported scale. The PGIS is a 1-item questionnaire designed to assess participant's impression of disease severity using a 5-point scale ranging from 1 to 5, where 1=none, 2=mild, 3=moderate, 4=severe, 5=very severe. Higher scores indicated greater severity. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: as for outcome 10
Population: Analysis was performed on Part B-FAS. Here, 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that none of participants were available for assessment at the specified timepoints. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]).
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
Participants
  Week 39 - None: number analyzed (Participants) | 17 | 17
  Week 39 - None | 7 | 5
  Week 39 - Mild: number analyzed (Participants) | 17 | 17
  Week 39 - Mild | 8 | 7
  Week 39 - Moderate: number analyzed (Participants) | 17 | 17
  Week 39 - Moderate | 1 | 5
  Week 39 - Severe: number analyzed (Participants) | 17 | 17
  Week 39 - Severe | 1 | 0
  Week 39 - Very Severe: number analyzed (Participants) | 17 | 17
  Week 39 - Very Severe | 0 | 0
  Week 51 - None: number analyzed (Participants) | 15 | 16
  Week 51 - None | 5 | 4
  Week 51 - Mild: number analyzed (Participants) | 15 | 16
  Week 51 - Mild | 8 | 7
  Week 51 - Moderate: number analyzed (Participants) | 15 | 16
  Week 51 - Moderate | 2 | 5
  Week 51 - Severe: number analyzed (Participants) | 15 | 16
  Week 51 - Severe | 0 | 0
  Week 51 - Very Severe: number analyzed (Participants) | 15 | 16
  Week 51 - Very Severe | 0 | 0
  Week 63 - None: number analyzed (Participants) | 17 | 16
  Week 63 - None | 6 | 4
  Week 63 - Mild: number analyzed (Participants) | 17 | 16
  Week 63 - Mild | 8 | 7
  Week 63 - Moderate: number analyzed (Participants) | 17 | 16
  Week 63 - Moderate | 3 | 5
  Week 63 - Severe: number analyzed (Participants) | 17 | 16
  Week 63 - Severe | 0 | 0
  Week 63 - Very Severe: number analyzed (Participants) | 17 | 16
  Week 63 - Very Severe | 0 | 0
  Week 75 - None: number analyzed (Participants) | 13 | 15
  Week 75 - None | 5 | 6
  Week 75 - Mild: number analyzed (Participants) | 13 | 15
  Week 75 - Mild | 6 | 6
  Week 75 - Moderate: number analyzed (Participants) | 13 | 15
  Week 75 - Moderate | 2 | 3
  Week 75 - Severe: number analyzed (Participants) | 13 | 15
  Week 75 - Severe | 0 | 0
  Week 75 - Very Severe: number analyzed (Participants) | 13 | 15
  Week 75 - Very Severe | 0 | 0
  Week 87 - None: number analyzed (Participants) | 13 | 15
  Week 87 - None | 6 | 7
  Week 87 - Mild: number analyzed (Participants) | 13 | 15
  Week 87 - Mild | 5 | 4
  Week 87 - Moderate: number analyzed (Participants) | 13 | 15
  Week 87 - Moderate | 1 | 3
  Week 87 - Severe: number analyzed (Participants) | 13 | 15
  Week 87 - Severe | 1 | 1
  Week 87 - Very Severe: number analyzed (Participants) | 13 | 15
  Week 87 - Very Severe | 0 | 0
  Week 99 - None: number analyzed (Participants) | 11 | 13
  Week 99 - None | 5 | 8
  Week 99 - Mild: number analyzed (Participants) | 11 | 13
  Week 99 - Mild | 5 | 3
  Week 99 - Moderate: number analyzed (Participants) | 11 | 13
  Week 99 - Moderate | 1 | 2
  Week 99 - Severe: number analyzed (Participants) | 11 | 13
  Week 99 - Severe | 0 | 0
  Week 99 - Very Severe: number analyzed (Participants) | 11 | 13
  Week 99 - Very Severe | 0 | 0
  Week 111 - None: number analyzed (Participants) | 11 | 12
  Week 111 - None | 5 | 7
  Week 111 - Mild: number analyzed (Participants) | 11 | 12
  Week 111 - Mild | 4 | 3
  Week 111 - Moderate: number analyzed (Participants) | 11 | 12
  Week 111 - Moderate | 2 | 2
  Week 111 - Severe: number analyzed (Participants) | 11 | 12
  Week 111 - Severe | 0 | 0
  Week 111 - Very Severe: number analyzed (Participants) | 11 | 12
  Week 111 - Very Severe | 0 | 0
  Week 123 - None: number analyzed (Participants) | 9 | 9
  Week 123 - None | 2 | 5
  Week 123 - Mild: number analyzed (Participants) | 9 | 9
  Week 123 - Mild | 6 | 2
  Week 123 - Moderate: number analyzed (Participants) | 9 | 9
  Week 123 - Moderate | 1 | 2
  Week 123 - Severe: number analyzed (Participants) | 9 | 9
  Week 123 - Severe | 0 | 0
  Week 123 - Very Severe: number analyzed (Participants) | 9 | 9
  Week 123 - Very Severe | 0 | 0
  Week 135 - None: number analyzed (Participants) | 5 | 5
  Week 135 - None | 0 | 2
  Week 135 - Mild: number analyzed (Participants) | 5 | 5
  Week 135 - Mild | 3 | 1
  Week 135 - Moderate: number analyzed (Participants) | 5 | 5
  Week 135 - Moderate | 2 | 2
  Week 135 - Severe: number analyzed (Participants) | 5 | 5
  Week 135 - Severe | 0 | 0
  Week 135 - Very Severe: number analyzed (Participants) | 5 | 5
  Week 135 - Very Severe | 0 | 0
  Week 147 - None: number analyzed (Participants) | 2 | 2
  Week 147 - None | 0 | 1
  Week 147 - Mild: number analyzed (Participants) | 2 | 2
  Week 147 - Mild | 1 | 0
  Week 147 - Moderate: number analyzed (Participants) | 2 | 2
  Week 147 - Moderate | 1 | 1
  Week 147 - Severe: number analyzed (Participants) | 2 | 2
  Week 147 - Severe | 0 | 0
  Week 147 - Very Severe: number analyzed (Participants) | 2 | 2
  Week 147 - Very Severe | 0 | 0
  Week 159 - None: number analyzed (Participants) | 1 | 1
  Week 159 - None | 0 | 0
  Week 159 - Mild: number analyzed (Participants) | 1 | 1
  Week 159 - Mild | 0 | 0
  Week 159 - Moderate: number analyzed (Participants) | 1 | 1
  Week 159 - Moderate | 1 | 1
  Week 159 - Severe: number analyzed (Participants) | 1 | 1
  Week 159 - Severe | 0 | 0
  Week 159 - Very Severe: number analyzed (Participants) | 1 | 1
  Week 159 - Very Severe | 0 | 0
  Week 171 - None: number analyzed (Participants) | 1 | 0
  Week 171 - None | 0 | 0
  Week 171 - Mild: number analyzed (Participants) | 1 | 0
  Week 171 - Mild | 1 | 0
  Week 171 - Moderate: number analyzed (Participants) | 1 | 0
  Week 171 - Moderate | 0 | 0
  Week 171 - Severe: number analyzed (Participants) | 1 | 0
  Week 171 - Severe | 0 | 0
  Week 171 - Very Severe: number analyzed (Participants) | 1 | 0
  Week 171 - Very Severe | 0 | 0
  ET/SFU - None: number analyzed (Participants) | 19 | 18
  ET/SFU - None | 2 | 4
  ET/SFU - Mild: number analyzed (Participants) | 19 | 18
  ET/SFU - Mild | 5 | 3
  ET/SFU - Moderate: number analyzed (Participants) | 19 | 18
  ET/SFU - Moderate | 7 | 5
  ET/SFU - Severe: number analyzed (Participants) | 19 | 18
  ET/SFU - Severe | 3 | 5
  ET/SFU - Very Severe: number analyzed (Participants) | 19 | 18
  ET/SFU - Very Severe | 2 | 1

14. Secondary Outcome: Part B: Number of Participants With Response to Participant's Global Impression of Change (PGIC) Questionnaire at Each Specified Time Points
Description: PGIC is a self-administered questionnaire to evaluate the improvement or worsening compared to the start of the study. PGIC was assessed on a 7-point Likert scale ranged from 1 (greatly improved) to 7 (greatly worsened). Categories were defined based on the PGIC scores as follows: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse and 7=very much worsen. Higher scores indicated greater severity. ET visit/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: as for outcome 10
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
Participants
  Week 39 - Very much improved: number analyzed (Participants) | 17 | 16
  Week 39 - Very much improved | 4 | 3
  Week 39 - Much improved: number analyzed (Participants) | 17 | 16
  Week 39 - Much improved | 8 | 6
  Week 39 - Minimally improved: number analyzed (Participants) | 17 | 16
  Week 39 - Minimally improved | 2 | 6
  Week 39 - No Change: number analyzed (Participants) | 17 | 16
  Week 39 - No Change | 2 | 1
  Week 39 - Minimally worse: number analyzed (Participants) | 17 | 16
  Week 39 - Minimally worse | 1 | 0
  Week 39 - Much worse: number analyzed (Participants) | 17 | 16
  Week 39 - Much worse | 0 | 0
  Week 39 - Very much worse: number analyzed (Participants) | 17 | 16
  Week 39 - Very much worse | 0 | 0
  Week 51 - Very much improved: number analyzed (Participants) | 15 | 16
  Week 51 - Very much improved | 5 | 3
  Week 51 - Much improved: number analyzed (Participants) | 15 | 16
  Week 51 - Much improved | 3 | 6
  Week 51 - Minimally improved: number analyzed (Participants) | 15 | 16
  Week 51 - Minimally improved | 2 | 4
  Week 51 - No Change: number analyzed (Participants) | 15 | 16
  Week 51 - No Change | 5 | 2
  Week 51 - Minimally worse: number analyzed (Participants) | 15 | 16
  Week 51 - Minimally worse | 0 | 0
  Week 51 - Much worse: number analyzed (Participants) | 15 | 16
  Week 51 - Much worse | 0 | 1
  Week 51 - Very much worse: number analyzed (Participants) | 15 | 16
  Week 51 - Very much worse | 0 | 0
  Week 63 - Very much improved: number analyzed (Participants) | 17 | 16
  Week 63 - Very much improved | 5 | 3
  Week 63 - Much improved: number analyzed (Participants) | 17 | 16
  Week 63 - Much improved | 8 | 4
  Week 63 - Minimally improved: number analyzed (Participants) | 17 | 16
  Week 63 - Minimally improved | 0 | 5
  Week 63 - No change: number analyzed (Participants) | 17 | 16
  Week 63 - No change | 4 | 3
  Week 63 - Minimally worse: number analyzed (Participants) | 17 | 16
  Week 63 - Minimally worse | 0 | 0
  Week 63 - Much worse: number analyzed (Participants) | 17 | 16
  Week 63 - Much worse | 0 | 1
  Week 63 - Very much worse: number analyzed (Participants) | 17 | 16
  Week 63 - Very much worse | 0 | 0
  Week 75 - Very much improved: number analyzed (Participants) | 13 | 15
  Week 75 - Very much improved | 6 | 6
  Week 75 - Much improved: number analyzed (Participants) | 13 | 15
  Week 75 - Much improved | 2 | 3
  Week 75 - Minimally improved: number analyzed (Participants) | 13 | 15
  Week 75 - Minimally improved | 1 | 5
  Week 75 - No Change: number analyzed (Participants) | 13 | 15
  Week 75 - No Change | 4 | 1
  Week 75 - Minimally worse: number analyzed (Participants) | 13 | 15
  Week 75 - Minimally worse | 0 | 0
  Week 75 - Much worse: number analyzed (Participants) | 13 | 15
  Week 75 - Much worse | 0 | 0
  Week 75 - Very much worse: number analyzed (Participants) | 13 | 15
  Week 75 - Very much worse | 0 | 0
  Week 87 - Very much improved: number analyzed (Participants) | 13 | 15
  Week 87 - Very much improved | 7 | 7
  Week 87 - Much improved: number analyzed (Participants) | 13 | 15
  Week 87 - Much improved | 0 | 3
  Week 87 - Minimally improved: number analyzed (Participants) | 13 | 15
  Week 87 - Minimally improved | 2 | 1
  Week 87 - No Change: number analyzed (Participants) | 13 | 15
  Week 87 - No Change | 2 | 3
  Week 87 - Minimally worse: number analyzed (Participants) | 13 | 15
  Week 87 - Minimally worse | 1 | 1
  Week 87 - Much worse: number analyzed (Participants) | 13 | 15
  Week 87 - Much worse | 1 | 0
  Week 87 - Very much worse: number analyzed (Participants) | 13 | 15
  Week 87 - Very much worse | 0 | 0
  Week 99 - Very much improved: number analyzed (Participants) | 11 | 13
  Week 99 - Very much improved | 3 | 8
  Week 99 - Much improved: number analyzed (Participants) | 11 | 13
  Week 99 - Much improved | 3 | 2
  Week 99 - Minimally improved: number analyzed (Participants) | 11 | 13
  Week 99 - Minimally improved | 1 | 3
  Week 99 - No change: number analyzed (Participants) | 11 | 13
  Week 99 - No change | 3 | 0
  Week 99 - Minimally worse: number analyzed (Participants) | 11 | 13
  Week 99 - Minimally worse | 1 | 0
  Week 99 - Much worse: number analyzed (Participants) | 11 | 13
  Week 99 - Much worse | 0 | 0
  Week 99 - Very much worse: number analyzed (Participants) | 11 | 13
  Week 99 - Very much worse | 0 | 0
  Week 111 - Very much improved: number analyzed (Participants) | 11 | 12
  Week 111 - Very much improved | 3 | 6
  Week 111 - Much improved: number analyzed (Participants) | 11 | 12
  Week 111 - Much improved | 5 | 4
  Week 111 - Minimally improved: number analyzed (Participants) | 11 | 12
  Week 111 - Minimally improved | 1 | 1
  Week 111 - No Change: number analyzed (Participants) | 11 | 12
  Week 111 - No Change | 2 | 1
  Week 111 - Minimally worse: number analyzed (Participants) | 11 | 12
  Week 111 - Minimally worse | 0 | 0
  Week 111 - Much worse: number analyzed (Participants) | 11 | 12
  Week 111 - Much worse | 0 | 0
  Week 111 - Very much worse: number analyzed (Participants) | 11 | 12
  Week 111 - Very much worse | 0 | 0
  Week 123 - Very much improved: number analyzed (Participants) | 9 | 9
  Week 123 - Very much improved | 3 | 4
  Week 123 - Much improved: number analyzed (Participants) | 9 | 9
  Week 123 - Much improved | 3 | 3
  Week 123 - Minimally improved: number analyzed (Participants) | 9 | 9
  Week 123 - Minimally improved | 2 | 1
  Week 123 - No Change: number analyzed (Participants) | 9 | 9
  Week 123 - No Change | 1 | 1
  Week 123 - Minimally worse: number analyzed (Participants) | 9 | 9
  Week 123 - Minimally worse | 0 | 0
  Week 123 - Much worse: number analyzed (Participants) | 9 | 9
  Week 123 - Much worse | 0 | 0
  Week 123 - Very much worse: number analyzed (Participants) | 9 | 9
  Week 123 - Very much worse | 0 | 0
  Week 135 - Very much improved: number analyzed (Participants) | 5 | 5
  Week 135 - Very much improved | 2 | 2
  Week 135 - Much improved: number analyzed (Participants) | 5 | 5
  Week 135 - Much improved | 2 | 1
  Week 135 - Minimally improved: number analyzed (Participants) | 5 | 5
  Week 135 - Minimally improved | 0 | 1
  Week 135 - No Change: number analyzed (Participants) | 5 | 5
  Week 135 - No Change | 0 | 1
  Week 135 - Minimally worse: number analyzed (Participants) | 5 | 5
  Week 135 - Minimally worse | 1 | 0
  Week 135 - Much worse: number analyzed (Participants) | 5 | 5
  Week 135 - Much worse | 0 | 0
  Week 135 - Very much worse: number analyzed (Participants) | 5 | 5
  Week 135 - Very much worse | 0 | 0
  Week 147 - Very much improved: number analyzed (Participants) | 2 | 2
  Week 147 - Very much improved | 1 | 0
  Week 147 - Much improved: number analyzed (Participants) | 2 | 2
  Week 147 - Much improved | 0 | 1
  Week 147 - Minimally improved: number analyzed (Participants) | 2 | 2
  Week 147 - Minimally improved | 0 | 1
  Week 147 - No Change: number analyzed (Participants) | 2 | 2
  Week 147 - No Change | 1 | 0
  Week 147 - Minimally worse: number analyzed (Participants) | 2 | 2
  Week 147 - Minimally worse | 0 | 0
  Week 147 - Much worse: number analyzed (Participants) | 2 | 2
  Week 147 - Much worse | 0 | 0
  Week 147 - Very much worse: number analyzed (Participants) | 2 | 2
  Week 147 - Very much worse | 0 | 0
  Week 159 - Very much improved: number analyzed (Participants) | 1 | 1
  Week 159 - Very much improved | 1 | 0
  Week 159 - Much improved: number analyzed (Participants) | 1 | 1
  Week 159 - Much improved | 0 | 0
  Week 159 - Minimally improved: number analyzed (Participants) | 1 | 1
  Week 159 - Minimally improved | 0 | 1
  Week 159 - No Change: number analyzed (Participants) | 1 | 1
  Week 159 - No Change | 0 | 0
  Week 159 - Minimally worse: number analyzed (Participants) | 1 | 1
  Week 159 - Minimally worse | 0 | 0
  Week 159 - Much worse: number analyzed (Participants) | 1 | 1
  Week 159 - Much worse | 0 | 0
  Week 159 - Very much worse: number analyzed (Participants) | 1 | 1
  Week 159 - Very much worse | 0 | 0
  Week 171- Very much improved: number analyzed (Participants) | 1 | 0
  Week 171- Very much improved | 1 | 0
  Week 171- Much improved: number analyzed (Participants) | 1 | 0
  Week 171- Much improved | 0 | 0
  Week 171- Minimally improved: number analyzed (Participants) | 1 | 0
  Week 171- Minimally improved | 0 | 0
  Week 171- No Change: number analyzed (Participants) | 1 | 0
  Week 171- No Change | 0 | 0
  Week 171- Minimally worse: number analyzed (Participants) | 1 | 0
  Week 171- Minimally worse | 0 | 0
  Week 171- Much worse: number analyzed (Participants) | 1 | 0
  Week 171- Much worse | 0 | 0
  Week 171- Very much worse: number analyzed (Participants) | 1 | 0
  Week 171- Very much worse | 0 | 0
  ET/SFU Visit- Very much improved: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Very much improved | 3 | 3
  ET/SFU Visit- Much improved: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Much improved | 5 | 6
  ET/SFU Visit- Minimally improved: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Minimally improved | 4 | 1
  ET/SFU Visit- No Change: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- No Change | 3 | 3
  ET/SFU Visit- Minimally worse: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Minimally worse | 1 | 2
  ET/SFU Visit- Much worse: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Much worse | 3 | 3
  ET/SFU Visit- Very much worse: number analyzed (Participants) | 19 | 18
  ET/SFU Visit- Very much worse | 0 | 0

15. Secondary Outcome: Part B: Mean Change From Baseline in Lactate Dehydrogenase (LDH) Level at Each Specified Time Points
Description: Change from baseline (Week 0) in LDH levels at each specified time points (i.e., Week 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 81, 83, 85, 87, 89, 91, 93, 95, 97, 99, 101, 103, 105, 107,109, 111, 113, 115, 117, 119, 121,123, 125, 127,129,131,133,135,137,139,141,143,145,147, 149, 151,153,155,157,159,161,163,165,167,169, 171, 173, 175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184).
Time Frame: Baseline (Week 0), every 2 weeks starting from Week 27 till Week 175 and at ET/SFU visit (i.e., up to Week 184)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
units per liter
  Week 27 | -151.000 (184.640) | 0.650 (208.051)
  Week 29: number analyzed (Participants) | 18 | 19
  Week 29 | -115.944 (226.913) | 11.000 (222.383)
  Week 31: number analyzed (Participants) | 18 | 17
  Week 31 | -85.111 (247.506) | 38.882 (211.386)
  Week 33: number analyzed (Participants) | 17 | 16
  Week 33 | -66.176 (324.145) | 4.813 (203.939)
  Week 35: number analyzed (Participants) | 18 | 16
  Week 35 | -64.667 (261.431) | -19.313 (142.989)
  Week 37: number analyzed (Participants) | 16 | 17
  Week 37 | 4.438 (398.843) | 25.765 (219.679)
  Week 39: number analyzed (Participants) | 16 | 16
  Week 39 | -88.500 (271.941) | 27.313 (210.705)
  Week 41: number analyzed (Participants) | 18 | 17
  Week 41 | 23.778 (342.195) | -6.000 (173.810)
  Week 43: number analyzed (Participants) | 17 | 17
  Week 43 | -22.118 (310.381) | -21.706 (181.668)
  Week 45: number analyzed (Participants) | 17 | 18
  Week 45 | 26.529 (329.717) | -13.500 (190.460)
  Week 47: number analyzed (Participants) | 15 | 18
  Week 47 | -22.600 (302.511) | -24.944 (153.580)
  Week 49: number analyzed (Participants) | 16 | 18
  Week 49 | -29.250 (289.392) | 15.722 (193.630)
  Week 51: number analyzed (Participants) | 16 | 18
  Week 51 | -12.563 (290.489) | -9.556 (155.646)
  Week 53: number analyzed (Participants) | 16 | 17
  Week 53 | -16.938 (299.788) | 12.529 (206.642)
  Week 55: number analyzed (Participants) | 14 | 16
  Week 55 | -89.500 (219.634) | -11.250 (177.647)
  Week 57: number analyzed (Participants) | 15 | 16
  Week 57 | -78.200 (285.140) | 64.188 (266.395)
  Week 59: number analyzed (Participants) | 16 | 17
  Week 59 | -84.438 (220.376) | 31.647 (226.128)
  Week 61: number analyzed (Participants) | 17 | 17
  Week 61 | -74.353 (215.414) | 20.588 (263.984)
  Week 63: number analyzed (Participants) | 17 | 17
  Week 63 | -98.235 (185.259) | 38.059 (325.329)
  Week 65: number analyzed (Participants) | 16 | 15
  Week 65 | -97.438 (212.335) | -16.467 (246.765)
  Week 67: number analyzed (Participants) | 17 | 15
  Week 67 | -127.824 (192.148) | 29.667 (269.918)
  Week 69: number analyzed (Participants) | 16 | 16
  Week 69 | -113.625 (197.270) | 36.563 (303.550)
  Week 71: number analyzed (Participants) | 13 | 15
  Week 71 | -101.692 (320.348) | 4.067 (307.924)
  Week 73: number analyzed (Participants) | 14 | 16
  Week 73 | -174.500 (177.153) | 7.063 (245.723)
  Week 75: number analyzed (Participants) | 14 | 15
  Week 75 | -157.429 (184.525) | 7.067 (285.183)
  Week 77: number analyzed (Participants) | 14 | 15
  Week 77 | -142.857 (199.169) | -24.867 (291.754)
  Week 79: number analyzed (Participants) | 13 | 16
  Week 79 | -98.077 (271.632) | -20.063 (265.761)
  Week 81: number analyzed (Participants) | 13 | 15
  Week 81 | -127.846 (233.663) | 7.200 (219.952)
  Week 83: number analyzed (Participants) | 13 | 11
  Week 83 | -59.000 (346.917) | 8.818 (250.068)
  Week 85: number analyzed (Participants) | 13 | 15
  Week 85 | -72.000 (350.021) | 28.400 (282.626)
  Week 87: number analyzed (Participants) | 13 | 13
  Week 87 | -101.385 (285.590) | 83.385 (288.731)
  Week 89: number analyzed (Participants) | 12 | 12
  Week 89 | -78.667 (351.059) | 10.833 (323.647)
  Week 91: number analyzed (Participants) | 9 | 13
  Week 91 | -143.000 (273.540) | 0.846 (288.451)
  Week 93: number analyzed (Participants) | 10 | 11
  Week 93 | -133.500 (254.332) | 10.818 (268.308)
  Week 95: number analyzed (Participants) | 11 | 13
  Week 95 | -59.364 (368.708) | 18.231 (241.354)
  Week 97: number analyzed (Participants) | 11 | 10
  Week 97 | -53.364 (343.820) | -38.500 (188.403)
  Week 99: number analyzed (Participants) | 11 | 12
  Week 99 | -80.909 (312.405) | -12.917 (183.844)
  Week 101: number analyzed (Participants) | 11 | 11
  Week 101 | -90.273 (293.680) | -17.182 (249.134)
  Week 103: number analyzed (Participants) | 11 | 13
  Week 103 | -50.273 (331.072) | 5.692 (211.233)
  Week 105: number analyzed (Participants) | 11 | 12
  Week 105 | -96.455 (276.907) | -34.250 (147.738)
  Week 107: number analyzed (Participants) | 11 | 13
  Week 107 | -28.091 (354.244) | 20.769 (222.772)
  Week 109: number analyzed (Participants) | 11 | 11
  Week 109 | -50.727 (335.078) | -2.000 (243.243)
  Week 111: number analyzed (Participants) | 10 | 12
  Week 111 | -83.000 (303.258) | -5.583 (219.850)
  Week 113: number analyzed (Participants) | 10 | 12
  Week 113 | -80.700 (319.283) | 0.667 (294.904)
  Week 115: number analyzed (Participants) | 10 | 10
  Week 115 | -109.500 (256.395) | 44.700 (295.946)
  Week 117: number analyzed (Participants) | 9 | 10
  Week 117 | -140.444 (280.944) | 12.700 (254.786)
  Week 119: number analyzed (Participants) | 9 | 10
  Week 119 | -149.556 (237.771) | -26.500 (274.168)
  Week 121: number analyzed (Participants) | 9 | 8
  Week 121 | -195.778 (225.978) | -42.375 (211.840)
  Week 123: number analyzed (Participants) | 9 | 9
  Week 123 | -185.000 (231.489) | 22.222 (278.037)
  Week 125: number analyzed (Participants) | 7 | 7
  Week 125 | -99.429 (285.513) | -85.143 (265.374)
  Week 127: number analyzed (Participants) | 7 | 8
  Week 127 | -154.714 (231.922) | -28.875 (312.483)
  Week 129: number analyzed (Participants) | 7 | 7
  Week 129 | -136.429 (234.954) | -18.571 (354.584)
  Week 131: number analyzed (Participants) | 6 | 6
  Week 131 | -120.833 (300.454) | -2.000 (270.245)
  Week 133: number analyzed (Participants) | 5 | 4
  Week 133 | -179.000 (298.811) | -47.500 (367.639)
  Week 135: number analyzed (Participants) | 5 | 5
  Week 135 | -211.800 (265.438) | 58.000 (449.233)
  Week 137: number analyzed (Participants) | 4 | 2
  Week 137 | -252.500 (264.591) | 46.500 (768.625)
  Week 139: number analyzed (Participants) | 5 | 3
  Week 139 | -181.800 (284.966) | -48.667 (373.339)
  Week 141: number analyzed (Participants) | 3 | 3
  Week 141 | -259.667 (362.136) | 30.667 (372.889)
  Week 143: number analyzed (Participants) | 4 | 2
  Week 143 | -160.250 (357.021) | -7.500 (21.920)
  Week 145: number analyzed (Participants) | 2 | 2
  Week 145 | -340.500 (458.912) | 290.000 (562.857)
  Week 147: number analyzed (Participants) | 3 | 2
  Week 147 | -248.667 (355.136) | 311.000 (547.301)
  Week 149: number analyzed (Participants) | 1 | 2
  Week 149 | -78.000 | 116.000 (175.362)
  Week 151: number analyzed (Participants) | 2 | 1
  Week 151 | 58.000 (32.527) | 295.000
  Week 153: number analyzed (Participants) | 1 | 1
  Week 153 | 7.000 | 75.000
  Week 155: number analyzed (Participants) | 1 | 0
  Week 155 | -50.000 |
  Week 157: number analyzed (Participants) | 1 | 1
  Week 157 | -50.000 | 369.000
  Week 159: number analyzed (Participants) | 1 | 1
  Week 159 | -155.000 | 365.000
  Week 161: number analyzed (Participants) | 1 | 0
  Week 161 | -175.000 |
  Week 163: number analyzed (Participants) | 1 | 1
  Week 163 | -149.000 | 782.000
  Week 165: number analyzed (Participants) | 1 | 0
  Week 165 | -155.000 |
  Week 167: number analyzed (Participants) | 1 | 0
  Week 167 | -162.000 |
  Week 169: number analyzed (Participants) | 1 | 0
  Week 169 | -180.000 |
  Week 171: number analyzed (Participants) | 1 | 0
  Week 171 | -167.000 |
  Week 173: number analyzed (Participants) | 1 | 0
  Week 173 | -171.000 |
  Week 175: number analyzed (Participants) | 1 | 0
  Week 175 | -121.000 |
  ET/SFU Visit: number analyzed (Participants) | 16 | 17
  ET/SFU Visit | -2.500 (195.967) | -11.706 (206.321)

16. Secondary Outcome: Part B: Number of Blood Transfusions Per Participant
Description: A participant was to receive a transfusion if his or her Hgb level met either of the following criteria: Hgb was <9 g/dL and the participant had symptoms of anemia or Hgb was <7 g/dL and the participant was asymptomatic.
Time Frame: From Week 27 up to 149 weeks of treatment (i.e., up to Week 176)
Population: Analysis was performed on Part B-FAS. Data for this outcome measure was planned to be collected and analyzed for combined population of BIVV009 (i.e., all participants who received BIVV009 [either 6.5 g or 7.5 g]).
Measure: Mean (Standard Deviation); unit: blood transfusions per participant
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
blood transfusions per participant | 0.4 (0.8) | 0.3 (0.4)

17. Secondary Outcome: Part B: Mean Change From Baseline in Haptoglobin Values at Each Specified Time Points
Description: Change from baseline (Week 0) in haptoglobin values at each specified time points (i.e., Week 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, 51, 53, 55, 57, 59, 61, 63, 65, 67, 69, 71, 73, 75, 77, 79, 81, 83, 85, 87, 89, 91, 93, 95, 97,99,101,103, 105, 107,109, 111,113,115,117,119, 121,123, 125, 127, 129,131,133,135,137,139,141,143, 145,147,149,151,153,155,157,159, 161,163,165,167,169,171,173,175 and ET/SFU Visit) is reported in this outcome measure. Baseline was defined as the last non-missing value prior to the first administration of study drug in Part A. ET/SFU visit was 9 weeks after administration of last dose (i.e., up to Week 184). Haptoglobin values <0.2 were imputed as 0.2.
Time Frame: Baseline (Week 0), every 2 weeks starting from Week 27 till Week 175 and at ET/SFU visit (i.e., up to Week 184)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
grams per liter
  Week 27: number analyzed (Participants) | 19 | 19
  Week 27 | 0.219 (0.380) | 0.082 (0.197)
  Week 29: number analyzed (Participants) | 18 | 20
  Week 29 | 0.240 (0.317) | 0.182 (0.482)
  Week 31 | 0.183 (0.311) | 0.256 (0.516)
  Week 33: number analyzed (Participants) | 19 | 17
  Week 33 | 0.212 (0.423) | 0.229 (0.379)
  Week 35: number analyzed (Participants) | 18 | 19
  Week 35 | 0.207 (0.355) | 0.151 (0.280)
  Week 37: number analyzed (Participants) | 18 | 18
  Week 37 | 0.232 (0.419) | 0.187 (0.291)
  Week 39: number analyzed (Participants) | 16 | 16
  Week 39 | 0.213 (0.330) | 0.165 (0.295)
  Week 41: number analyzed (Participants) | 19 | 18
  Week 41 | 0.119 (0.238) | 0.082 (0.168)
  Week 43: number analyzed (Participants) | 18 | 18
  Week 43 | 0.100 (0.224) | 0.161 (0.234)
  Week 45: number analyzed (Participants) | 18 | 20
  Week 45 | 0.114 (0.205) | 0.189 (0.275)
  Week 47: number analyzed (Participants) | 15 | 20
  Week 47 | 0.135 (0.243) | 0.255 (0.416)
  Week 49: number analyzed (Participants) | 16 | 18
  Week 49 | 0.139 (0.205) | 0.172 (0.345)
  Week 51: number analyzed (Participants) | 15 | 17
  Week 51 | 0.083 (0.197) | 0.207 (0.369)
  Week 53: number analyzed (Participants) | 16 | 19
  Week 53 | 0.045 (0.137) | 0.122 (0.296)
  Week 55: number analyzed (Participants) | 17 | 18
  Week 55 | 0.149 (0.251) | 0.179 (0.343)
  Week 57: number analyzed (Participants) | 16 | 17
  Week 57 | 0.158 (0.234) | 0.158 (0.362)
  Week 59: number analyzed (Participants) | 17 | 17
  Week 59 | 0.132 (0.229) | 0.131 (0.306)
  Week 61: number analyzed (Participants) | 17 | 18
  Week 61 | 0.153 (0.286) | 0.184 (0.350)
  Week 63: number analyzed (Participants) | 17 | 17
  Week 63 | 0.202 (0.265) | 0.177 (0.357)
  Week 65: number analyzed (Participants) | 16 | 16
  Week 65 | 0.101 (0.232) | 0.198 (0.384)
  Week 67: number analyzed (Participants) | 17 | 16
  Week 67 | 0.178 (0.241) | 0.162 (0.363)
  Week 69: number analyzed (Participants) | 16 | 17
  Week 69 | 0.168 (0.255) | 0.169 (0.348)
  Week 71: number analyzed (Participants) | 14 | 15
  Week 71 | 0.220 (0.288) | 0.236 (0.388)
  Week 73: number analyzed (Participants) | 14 | 16
  Week 73 | 0.261 (0.335) | 0.174 (0.348)
  Week 75: number analyzed (Participants) | 15 | 16
  Week 75 | 0.275 (0.321) | 0.197 (0.362)
  Week 77: number analyzed (Participants) | 14 | 16
  Week 77 | 0.249 (0.374) | 0.232 (0.398)
  Week 79: number analyzed (Participants) | 14 | 16
  Week 79 | 0.299 (0.419) | 0.290 (0.464)
  Week 81: number analyzed (Participants) | 13 | 16
  Week 81 | 0.438 (0.463) | 0.207 (0.421)
  Week 83: number analyzed (Participants) | 14 | 13
  Week 83 | 0.297 (0.379) | 0.233 (0.394)
  Week 85: number analyzed (Participants) | 13 | 15
  Week 85 | 0.374 (0.374) | 0.266 (0.426)
  Week 87: number analyzed (Participants) | 12 | 13
  Week 87 | 0.334 (0.409) | 0.344 (0.471)
  Week 89: number analyzed (Participants) | 12 | 13
  Week 89 | 0.348 (0.482) | 0.198 (0.351)
  Week 91: number analyzed (Participants) | 11 | 12
  Week 91 | 0.313 (0.449) | 0.279 (0.449)
  Week 93: number analyzed (Participants) | 11 | 12
  Week 93 | 0.262 (0.383) | 0.178 (0.373)
  Week 95: number analyzed (Participants) | 11 | 13
  Week 95 | 0.263 (0.495) | 0.198 (0.414)
  Week 97: number analyzed (Participants) | 11 | 12
  Week 97 | 0.245 (0.306) | 0.210 (0.407)
  Week 99: number analyzed (Participants) | 11 | 13
  Week 99 | 0.266 (0.351) | 0.213 (0.370)
  Week 101: number analyzed (Participants) | 11 | 12
  Week 101 | 0.289 (0.289) | 0.207 (0.417)
  Week 103: number analyzed (Participants) | 11 | 13
  Week 103 | 0.219 (0.291) | 0.212 (0.389)
  Week 105: number analyzed (Participants) | 11 | 12
  Week 105 | 0.216 (0.291) | 0.174 (0.399)
  Week 107: number analyzed (Participants) | 11 | 13
  Week 107 | 0.182 (0.273) | 0.245 (0.459)
  Week 109: number analyzed (Participants) | 10 | 11
  Week 109 | 0.207 (0.311) | 0.254 (0.507)
  Week 111: number analyzed (Participants) | 11 | 12
  Week 111 | 0.282 (0.556) | 0.263 (0.459)
  Week 113: number analyzed (Participants) | 11 | 12
  Week 113 | 0.248 (0.366) | 0.335 (0.614)
  Week 115: number analyzed (Participants) | 10 | 11
  Week 115 | 0.324 (0.413) | 0.165 (0.432)
  Week 117: number analyzed (Participants) | 9 | 10
  Week 117 | 0.450 (0.492) | 0.181 (0.489)
  Week 119: number analyzed (Participants) | 9 | 10
  Week 119 | 0.348 (0.400) | 0.187 (0.404)
  Week 121: number analyzed (Participants) | 9 | 8
  Week 121 | 0.459 (0.414) | 0.174 (0.479)
  Week 123: number analyzed (Participants) | 9 | 9
  Week 123 | 0.350 (0.375) | 0.192 (0.512)
  Week 125: number analyzed (Participants) | 8 | 7
  Week 125 | 0.303 (0.425) | 0.114 (0.298)
  Week 127: number analyzed (Participants) | 7 | 8
  Week 127 | 0.309 (0.401) | 0.220 (0.420)
  Week 129: number analyzed (Participants) | 7 | 7
  Week 129 | 0.393 (0.506) | 0.191 (0.506)
  Week 131: number analyzed (Participants) | 6 | 5
  Week 131 | 0.480 (0.529) | 0.222 (0.430)
  Week 133: number analyzed (Participants) | 5 | 4
  Week 133 | 0.342 (0.469) | 0.125 (0.155)
  Week 135: number analyzed (Participants) | 5 | 5
  Week 135 | 0.454 (0.643) | 0.280 (0.425)
  Week 137: number analyzed (Participants) | 4 | 3
  Week 137 | 0.545 (0.631) | 0.070 (0.121)
  Week 139: number analyzed (Participants) | 5 | 3
  Week 139 | 0.494 (0.676) | 0.293 (0.508)
  Week 141: number analyzed (Participants) | 3 | 2
  Week 141 | 0.667 (0.583) | 0.025 (0.035)
  Week 143: number analyzed (Participants) | 4 | 3
  Week 143 | 0.513 (0.604) | 0.270 (0.292)
  Week 145: number analyzed (Participants) | 2 | 3
  Week 145 | 0.580 (0.820) | 0.130 (0.141)
  Week 147: number analyzed (Participants) | 3 | 2
  Week 147 | 0.400 (0.592) | 0.195 (0.276)
  Week 149: number analyzed (Participants) | 1 | 2
  Week 149 | 0.000 | 0.000 (0.000)
  Week 151: number analyzed (Participants) | 2 | 1
  Week 151 | 0.000 (0.000) | 0.000
  Week 153: number analyzed (Participants) | 1 | 1
  Week 153 | 0.000 | 0.000
  Week 155: number analyzed (Participants) | 1 | 1
  Week 155 | 0.000 | 0.000
  Week 157: number analyzed (Participants) | 1 | 1
  Week 157 | 0.000 | 0.000
  Week 159: number analyzed (Participants) | 1 | 1
  Week 159 | 0.000 | 0.000
  Week 161: number analyzed (Participants) | 1 | 1
  Week 161 | 0.180 | 0.000
  Week 163: number analyzed (Participants) | 1 | 1
  Week 163 | 0.000 | 0.000
  Week 165: number analyzed (Participants) | 1 | 0
  Week 165 | 0.000 |
  Week 167: number analyzed (Participants) | 1 | 0
  Week 167 | 0.000 |
  Week 169: number analyzed (Participants) | 1 | 0
  Week 169 | 0.000 |
  Week 171: number analyzed (Participants) | 1 | 0
  Week 171 | 0.000 |
  Week 173: number analyzed (Participants) | 1 | 0
  Week 173 | 0.000 |
  Week 175: number analyzed (Participants) | 1 | 0
  Week 175 | 0.000 |
  ET/SFU Visit: number analyzed (Participants) | 19 | 18
  ET/SFU Visit | 0.055 (0.200) | 0.181 (0.426)

18. Secondary Outcome: Part B: Number of Healthcare Visits by Type
Description: In this outcome measure, number of healthcare visits which included non-study healthcare resource utilization visit (consisted mainly of extra visits to the office of the study doctor, visit to a generalist doctor or visit to a specialist doctor), hospitalization visit and visit to hospital emergency is reported.
Time Frame: From Week 27 up to 149 weeks of treatment (i.e., up to Week 176)
Population: as for outcome 16
Measure: Number; unit: visits
Arm/Group | BIVV009/BIVV009 | Placebo/BIVV009
Number analyzed (Participants) | 19 | 20
visits
  Non-study healthcare resource utilization visits | 13 | 12
  Hospitalization | 3 | 1
  Visit to a hospital emergency room | 1 | 3

ADVERSE EVENTS:
Time Frame: Part A (both 6.5 g and 7.5 g cohorts): first dose (Day 0) up to Week 25; Part B, 6.5 g cohort: From first dose (Week 26) up to 149 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 184); Part B, 7.5 g cohort: From first dose (Week 26) up to 137 weeks of treatment + 9 weeks of follow-up (i.e., up to Week 172)
Description: Reported AEs and SAEs including fatal AEs were TEAEs that developed/worsened or became serious during on-treatment period. Analysis was performed on SAS.
Groups:
- Part A: BIVV009 6.5 g: Participants with primary CAD and body weight <75 kg and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of BIVV009 6.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
- Part A: BIVV009 7.5 g: Participants with primary CAD and body weight >=75 kg and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of BIVV009 7.5 g on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
- Part A: Placebo: Participants with primary CAD and without a recent history of blood transfusion during the last 6 months prior to enrollment in this study, received an IV infusion of placebo matched to BIVV009 on Day 0 and Day 7 and every 14 days thereafter in Part A up to Week 25.
Arm/Group | Part A: BIVV009 6.5 g | Part A: BIVV009 7.5 g | Part A: Placebo | Part B: BIVV009 6.5 g | Part B: BIVV009 7.5 g
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/5 | 0/20 | 1/32 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/5 | 0/20 | 6/32 | 1/7
Other Adverse Events (participants affected / at risk) | 16/17 | 5/5 | 3/20 | 28/32 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: BIVV009 6.5 g (N=17) | Part A: BIVV009 7.5 g (N=5) | Part A: Placebo (N=20) | Part B: BIVV009 6.5 g (N=32) | Part B: BIVV009 7.5 g (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polycystic Liver Disease (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Immunoglobulin M Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Venous Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Raynaud's Phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: BIVV009 6.5 g (N=17) | Part A: BIVV009 7.5 g (N=5) | Part A: Placebo (N=20) | Part B: BIVV009 6.5 g (N=32) | Part B: BIVV009 7.5 g (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 9 (11) | 2 (3)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Angular Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (4) | 0 (0) | 6 (13) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Faeces Discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 2 (2)
Catheter Site Dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (2) | 0 (0) | 7 (7) | 5 (10)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 1 (1)
Vaccination Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination Site Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vaccination Site Rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 5 (9) | 2 (3)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (4) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal Skin Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulval Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (3)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaccination Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Blood Immunoglobulin M Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood Urine Present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 6 (7) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bone Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (7) | 1 (1) | 0 (0) | 4 (9) | 2 (5)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phantom Limb Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Kink (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depressed Mood (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 4 (8) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Renal Cyst (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Calcifications (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyanosis (Vascular disorders) | 4 (10) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Extremity Necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (7) | 1 (1) | 0 (0) | 5 (7) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poor Venous Access (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Raynaud's Phenomenon (Vascular disorders) | 3 (4) | 1 (2) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03347422/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT03347422/SAP_001.pdf